CLINICAL TRIAL: NCT03174808
Title: Mindfulness Interventions and Cutaneous T Cell Lymphoma (CTCL)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI unexpectedly passed away, study closed.
Sponsor: Yale University (Other)
Collaborators: The Wallace Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000020161
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Anxiety; Quality of Life
Keywords: cutaneous T-cell lymphoma
MeSH Terms: conditions — Anxiety Disorders; Lymphoma, T-Cell, Cutaneous | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Stress Reduction (MBSR) (Experimental): Participants will attend group sessions led by an instructor experienced in MBSR in an academic setting.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Participants will attend weekly 2.5-hour group sessions (of 10-14 persons) based on the standard MBSR protocol.

SUMMARY:
The primary objective is to assess the feasibly, adherence, and effects of mindfulness-based stress reduction (MBSR) on anxiety and health-related quality of life in adult patients with cutaneous T-cell lymphoma at the Yale Cancer Center/Smilow Cancer Hospital.

Participants will attend group sessions led by an instructor experienced in MBSR in an academic setting. The mindfulness meditation group sessions will take place at the Smilow Cancer Center at the Yale New-Haven Hospital.

DETAILED DESCRIPTION:
Participants will attend weekly 2.5-hour group sessions (of 10-14 persons) based on the standard mindfulness-based stress reduction (MBSR) protocol. Participants will be assigned home practice based on the MBSR protocol, and will be given audio recordings (MP3) to accompany and instruct in home practice.

Eligible participants will attend weekly group sessions for 8 weeks and will be assessed at baseline, following cessation of the intervention (8-weeks), and 16 weeks. Outcomes will be assessed at baseline, 8 weeks, and 16 weeks. Extended effects of the intervention will be assessed at 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Identified with lymphoma through the Yale Cancer Center Hematology Clinic.
* Access to mobile telephone/smartphone with text messaging plan in order to receive survey questions.
* Current CTCL patients in Dr. Foss's practice at the Yale Cancer Center.

Exclusion Criteria:

* Current regular mindfulness meditation activity (weekly or more frequent practice of self-defined meditation, formalized relaxation techniques, tai chi, and meditative yoga).
* Inability or unwillingness to give consent.
* Serious illness (including mental illness/psychopathology) within 90 days prior to screening, including hospitalization for chronic disease. Determination of 'serious' will be made by PI and research team. For example, unstable asthma, cancers (except non-melanoma skin cancer and CTCL), and schizophrenia will be considered 'serious,' while stable asthma, allergic rhinitis, esophageal reflux, generalized anxiety disorder, or attention deficit disorder will not be considered 'serious.
* Active participation (weekly or more often) in a cancer or chronic disease support group.
* Active substance abusers.
* Current suicidal ideation, operationally defined as affirmative responses on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Feasibility | 16 weeks
  Feasibility of the intervention will be assessed by the proportion of eligible patients attend the majority of the MBSR sessions (5 or more), and complete week-8 and week-16 assessments.
Adherence | 16 weeks
  Adherence will be tracked by assessing the actual amount of home practice in minutes per week using weekly practice logs and/or SMS (short message service)/text messaging. Adherence will be quantitatively assessed through tallying home practice time and number of intervention visits attended.

SECONDARY OUTCOMES:
Stress | baseline, 8 weeks, and 16 weeks
  The Perceived Stress Scale (PSS) has been used in past Mindfulness treatment studies. The PSS is a 14-item scale that assesses perceived stress of life situations in adolescents and adults. Items are scored on a 5-point scale (0=never to 4=very often) (e.g., 'How often have you been upset because of something that happened unexpectedly?). Higher total scores indicate greater levels of perceived stress.
Quality of Life | baseline, 8 weeks, and 16 weeks
  The Functional Assessment of Cancer Therapy-General (FACT-G) is a cancer-focused measure of quality of life and well-being. It is a standard assessment at the Yale Survivorship clinic. It includes 27 items and encompasses 4 different indices of well-being: physical, social/family, emotional, and functional well-being and has been used to evaluate cancer-related QOL in many studies.

OTHER OUTCOMES:
Depression | baseline, 8 weeks, and 16 weeks
  The Hospital Anxiety and Depression Scale (HADS) has been used to measure levels of anxiety and depression that a patient is experiencing. The HADS has fourteen items, seven of which relate to anxiety and other seven of which related to depression. Each item is scored on a 0-3 scale. Higher total scores indicate greater levels of perceived anxiety/depression.
Anxiety | baseline, 8 weeks, and 16 weeks
  The Hospital Anxiety and Depression Scale (HADS) has been used to measure levels of anxiety and depression that a patient is experiencing. The HADS has fourteen items, seven of which relate to anxiety and other seven of which related to depression. Each item is scored on a 0-3 scale. Higher total scores indicate greater levels of perceived anxiety/depression.
Healing | baseline, 8 weeks, and 16 weeks
  The Healing Encounters and Attitudes Lists (HEAL) questionnaires have been used to measure the nonspecific factors in healing process including patient-provider connection, treatment expectancy, healthcare environment, positive outlook, spirituality and attitude towards complementary and alternative medicine. The HEAL item banks comprise six subscales, each of which has 6-7 questions. Each item is scored on a 1-5 scale. The HEAL measures have been well validated in integrative medicine research.
Effect of Skin Disease | baseline, 8 weeks, and 16 weeks
  The Skindex-29 profiles are a 29-item measure that assesses the symptomatic, emotional, and functional effects of skin diseases on quality of life. It is widely used in patients with nonmelanoma skin cancer including CTCL. Items are scored based on how often (Never, Rarely, Sometimes, Often, All the time) during the previous four weeks the patient experienced the effect described in each item. All responses are transformed to a linear scale of 100, varying from 0 (no effect) to 100 (effect experienced all the time).
Client Credibility | week 1
  The Client Credibility Questionnaire (CCQ) will be used to assess subject expectations and beliefs about the mindfulness program at baseline using a questionnaire modeled after the methods of Sherman et al. The CCQ will be administered to all subjects at the end of the first MBSR class, after the outline and rationale of the intervention has been presented. Subjects will be asked to make ratings using an 8-point Likert scale (0= not at all to 8=very much) about: (1) how logical the program seems; (2) how confident they are the program will be successful in reducing symptoms; and (3) how confident they would be in recommending the program to a friend.
Suicide Severity | screening/baseline
  Columbia-Suicide Severity Rating Scale (C-SSRS) is a 2-item, self-report questionnaire that includes items suicidal ideations in the past week and the past year. Questions include: (1) Have you wished you were dead or wished you could go to sleep and not wake up? and (2) Have you actually had any thoughts of killing yourself? Any positive (yes) responses during the past week are immediately referred to Yale-New Haven Children's Hospital.
Disease Progress | baseline, 8 weeks, and 16 weeks
  The Eastern Cooperative Oncology Group (ECOG) assessment will be used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. ECOG is graded from 0 to 5.
  0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; 5 = Dead .

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Shapiro, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center/Smilow, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided